CLINICAL TRIAL: NCT01804452
Title: Observational Longitudinal Study of Magnetic Resonance Imaging, Specimen Biomarkers, and Clinical Progression in Progressive Supranuclear Palsy and Corticobasal Degeneration
Brief Title: 4 Repeat Tauopathy Neuroimaging Initiative
Acronym: 4RTNI
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4RTNI; R01AG031278 (NIH)
Record Dates: First submitted 2013-01-18; First posted 2013-03-05 (Estimated); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Progressive Supranuclear Palsy; Corticobasal Degeneration
Keywords: Progressive Supranuclear Palsy; Corticobasal Degeneration; Biomarker; Neuroimaging; MRI; Tau; Oculomotor
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Corticobasal Degeneration; Pick Disease of the Brain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, urine, cell lines and cerebrospinal fluid will be retained by study investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with a diagnosis of PSP or CBD
  Interventions: Other: Observational Study

INTERVENTIONS:
Other: Observational Study

SUMMARY:
The purpose of this study is to evaluate several different tests, including brain imaging, eye movement testing, body fluid samples, measurements of memory and other thinking abilities, and measures of functional independence in the hope that this information can be used to guide diagnosis and treatment of PSP and CBD in the future. Recent advances in our understanding of the biological causes of these diseases offer hope for new treatments. As such treatments are developed, sensitive and specific biological measurements (biomarkers) will be needed to provide precise and direct measures of the state of the brain, which will improve the statistical power of clinical trials. Brain imaging with Magnetic Resonance Imaging (MRI) has previously been used to measure disease-related changes in the brain. The goal of this study is to identify the best methods of analysis (including eye movements, imaging, and behavioral measures) for tracking PSP and CBD over time. In addition, certain biomarkers in the blood and cerebrospinal fluid might also be useful for following these diseases over time. This study will examine the value of blood and CSF biomarkers relative to brain imaging and functional measures.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Progressive Supranuclear Palsy or Corticobasal Degeneration
* Must have a reliable study partner who has frequent contact with the subject
* Willing and able to undergo testing procedures

Exclusion Criteria:

* Significant neurological disease other than PSP or CBD
* Presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of PSP or CBD
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2011-01-10 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Progressive Supranuclear Palsy Rating Scale | Baseline, 6 months and 1 year
  Change from baseline

SECONDARY OUTCOMES:
Eye movement function | Baseline, 6 months and 1 year
  Change from baseline
Brain volume on MRI | Baseline, 6 months and 1 year
  Change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Boxer, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - John Hopkins University, Baltimore, Maryland

REFERENCES:
- [Background] Lee SE, Rabinovici GD, Mayo MC, Wilson SM, Seeley WW, DeArmond SJ, Huang EJ, Trojanowski JQ, Growdon ME, Jang JY, Sidhu M, See TM, Karydas AM, Gorno-Tempini ML, Boxer AL, Weiner MW, Geschwind MD, Rankin KP, Miller BL. Clinicopathological correlations in corticobasal degeneration. Ann Neurol. 2011 Aug;70(2):327-40. doi: 10.1002/ana.22424. PMID 21823158
- [Background] Coppola G, Chinnathambi S, Lee JJ, Dombroski BA, Baker MC, Soto-Ortolaza AI, Lee SE, Klein E, Huang AY, Sears R, Lane JR, Karydas AM, Kenet RO, Biernat J, Wang LS, Cotman CW, Decarli CS, Levey AI, Ringman JM, Mendez MF, Chui HC, Le Ber I, Brice A, Lupton MK, Preza E, Lovestone S, Powell J, Graff-Radford N, Petersen RC, Boeve BF, Lippa CF, Bigio EH, Mackenzie I, Finger E, Kertesz A, Caselli RJ, Gearing M, Juncos JL, Ghetti B, Spina S, Bordelon YM, Tourtellotte WW, Frosch MP, Vonsattel JP, Zarow C, Beach TG, Albin RL, Lieberman AP, Lee VM, Trojanowski JQ, Van Deerlin VM, Bird TD, Galasko DR, Masliah E, White CL, Troncoso JC, Hannequin D, Boxer AL, Geschwind MD, Kumar S, Mandelkow EM, Wszolek ZK, Uitti RJ, Dickson DW, Haines JL, Mayeux R, Pericak-Vance MA, Farrer LA; Alzheimer's Disease Genetics Consortium; Ross OA, Rademakers R, Schellenberg GD, Miller BL, Mandelkow E, Geschwind DH. Evidence for a role of the rare p.A152T variant in MAPT in increasing the risk for FTD-spectrum and Alzheimer's diseases. Hum Mol Genet. 2012 Aug 1;21(15):3500-12. doi: 10.1093/hmg/dds161. Epub 2012 May 3. PMID 22556362
- [Background] Garbutt S, Matlin A, Hellmuth J, Schenk AK, Johnson JK, Rosen H, Dean D, Kramer J, Neuhaus J, Miller BL, Lisberger SG, Boxer AL. Oculomotor function in frontotemporal lobar degeneration, related disorders and Alzheimer's disease. Brain. 2008 May;131(Pt 5):1268-81. doi: 10.1093/brain/awn047. Epub 2008 Mar 24. PMID 18362099
- [Background] Boxer AL, Geschwind MD, Belfor N, Gorno-Tempini ML, Schauer GF, Miller BL, Weiner MW, Rosen HJ. Patterns of brain atrophy that differentiate corticobasal degeneration syndrome from progressive supranuclear palsy. Arch Neurol. 2006 Jan;63(1):81-6. doi: 10.1001/archneur.63.1.81. PMID 16401739
- [Background] Belfor N, Amici S, Boxer AL, Kramer JH, Gorno-Tempini ML, Rosen HJ, Miller BL. Clinical and neuropsychological features of corticobasal degeneration. Mech Ageing Dev. 2006 Feb;127(2):203-7. doi: 10.1016/j.mad.2005.09.013. Epub 2005 Nov 28. PMID 16310834